CLINICAL TRIAL: NCT00199862
Title: A Pilot Study of Radioimmunodetection of 124-Iodine-labeled Humanized A33 Antibody (124I-huA33) in Patients With Colorectal Cancer
Brief Title: Safety Study of Radio-labeled huA33 Antibody in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-124
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Colorectal Tumor; COlorectal Carcinoma
Keywords: huA33; antibody; colorectal cancer; Iodine 124; 124I; 03-124
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Antibodies

ARMS (1):
- Radio-labeled huA33 Antibody (Experimental): Patients will receive a single I-V infusion of 4mCi-10mCi/10mg 124I-huA33 in 5-30 mL of 5% human serum albumin (HAS) in normal saline, over 5 minutes-4 hours. Patients will be studied with 124I-huA33 positron-emission tomography (PET) and ex-vivo quantitation of tumor uptake .
  Blood samples will be obtained for pharmacokinetic analysis at 5, 15, 60, and 120 minutes after completion of IV, on and before or after PET scanning on subsequent days.
  Surgery (or biopsy) will be scheduled to occur 8- 10 days after administration of 124I-huA33. The 8-10 day imaging session will be scheduled for the morning of surgery or biopsy, approximately 1-6 hours before the procedure.
  Interventions: Drug: Iodine-124 labeled humanized A33 (antibody)

INTERVENTIONS:
Drug: Iodine-124 labeled humanized A33 (antibody) — Patients will receive a single intravenous or intraarterial infusion of 10mg huA33, labeled with 4mCi-10mCi of 124I in 5-30ml of 5% HSA in normal saline (NS), over 5-10 minutes. On study days 2, 3, and/or 4 patients will have the option to receive up to 2g/kg of IVIG. Patients will be evaluated with 124I-huA33 positron-emission tomography (PET) with ex vivo quantitation of tumor uptake.

SUMMARY:
The purpose of this study is to determine whether our drug, 124I-huA33, can safely detect colorectal cancer.

DETAILED DESCRIPTION:
This is an open-label, pilot study of a single 4mCi-10mCi/10mg IV dose of 124I-huA33 in patients with colorectal cancer. Patients will be studied with 124I-huA33 positron-emission tomography (PET), and in the subset of patients scheduled for surgery, based on clinical indications, ex vivo quantitation of tumor uptake will also be performed. Patients will receive a single intravenous or intraarterial infusion of 4 mCi-10mCi /10mg 124I-huA33 in 5-30ml of 5% human serum albumin (HSA), over 5-10 minutes. Patient will either receive the 124I-huA33 intravenously (IV) or intraarterially (IA) to determine if there is an advantage of the IV vs the IA route. Following injection with 124I-huA33, on study days 2, 3, and/ or 4, patients will have the option to receive up to 2g/1kg of Immune Globulin (IVIG).

Blood samples will be obtained for pharmacokinetic analysis at 5, 15, 60, and 120 minutes after completion of IV or IA infusion, on day 2, 3, and/ or 4, and before and after the PET scan on the day of surgery or last imaging day (day 8 + 3). Patients scheduled for surgery will undergo a PET scan of the abdomen and pelvis 1-6 hours prior to surgery.

In those patients undergoing surgery, surgery (or biopsy) will be scheduled to occur day 8 (± 3 days) days after administration of 124I-huA33. Biopsy sites may include tumor, tumor bed, regional nodes, portal, suprapancreatic, celiac nodes and the retroperitoneum. Tumor and normal tissue obtained at surgery (or biopsy), and serum will be measured for estimation of percent-injected dose per gram of tumor, normal liver, and serum. Tissue samples will be obtained for autoradiography and immunohistochemistry as an additional assessment of tumor targeting.

Blood samples to determine immunogenicity will be taken at baseline and at 4 weeks.

Toxicity assessments will be made throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Primary or metastatic colorectal carcinoma, histologically confirmed at Memorial Sloan-Kettering Cancer Center (MSKCC).
* Patients must be candidates for clinically indicated surgery/biopsy for primary/metastatic colorectal cancer
* Expected survival of at least 3 months.
* Karnofsky performance status ≥ 70 (ECOG 0 or 1).
* The following laboratory results within the last 2 weeks prior to study day 1:

Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 75 x 109/L Serum bilirubin ≤ 2.5 mg/dL Serum creatinine ≤ 2.0 mg/dL White Blood Count (WBC) ≥ 3,000/mm3 Age ≥ 18 years. Children of all ages are not included as colon cancer is extremely rare in children.

* Women of childbearing potential with confirmed negative pregnancy test on the day of administration of study agent.
* Before any trial-specific procedures or treatment can be performed, the patient or patient's legally authorized guardian or representative must give witnessed written informed consent for participation in the tria

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III/IV).
* Active CNS tumor involvement. Previous treatment with A33 or its fragment and/or a positive test for huA33 HAHA.
* Lack of availability for immunological and clinical follow-up assessments.
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-02 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
To determine and quantify tumor uptake of radiolabeled antibody from measurements with: | Until end of study
PET imaging/Dosimetry | Until end of study
Autoradiographs - tumor or biopsy samples | Until end of study
Ex vivo radioactivity estimates - tumor, normal tissue and serum samples | Until end of study
Toxicity defined by NCI Common Toxicity Criteria | Until end of study

SECONDARY OUTCOMES:
Serum radioactivity, volume of distribution, and half-life following IV and IA 124I-huA33 | Until end of study
HAHA levels - measured by plasmon resonance surface (Biacore®) assay | Until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/